CLINICAL TRIAL: NCT06266793
Title: Comparison of Lumenis Pulse 120H Moses 2.0 Holmium Laser vs. Olympus Soltive Thulium Fiber Laser for Mini-percutaneous Nephrolithotomy
Brief Title: Comparison of Holmium Laser and Thulium Laser for Mini PCNL
Acronym: HOTLaser
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, David Sobel, Principal Investigator, MD, MaineHealth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2072488-2
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-02

CONDITIONS: Nephrolithiasis; Percutaneous Nephrolithotomy
Keywords: Laser; Holmium laser; Thulium fiber laser; PCNL; Nephrolithiasis; Percutaneous Nephrolithotomy
MeSH Terms: conditions — Nephrolithiasis | interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Holmium Laser (Active Comparator): Participants in this arm are randomized to be treated using the Lumenis Pulse 120H Moses 2.0 Holmium Laser
  Interventions: Device: Holmium Laser
- Thulium Laser (Active Comparator): Participants in this arm are randomized to be treated using the Olympus Soltive SuperPulsed Thulium Fiber Laser
  Interventions: Device: Thulium Laser

INTERVENTIONS:
Device: Holmium Laser — Assigned to be treated using the Lumenis Pulse 120H Moses 2.0 Holmium Laser.
  Arms: Holmium Laser
Device: Thulium Laser — Assigned to be treated using the Olympus Soltive Thulium SuperPulsed Fiber Laser
  Arms: Thulium Laser

SUMMARY:
This is a single institution, single surgeon, randomized controlled trial to evaluate the Boston Scientific Lumenis Pulse 120H Moses 2.0 holmium laser versus the Olympus Soltive Superpulsed thulium fiber laser (TFL) for medium-to-large stones in the mini PCNL setting.

DETAILED DESCRIPTION:
Multiple procedural modalities for treating nephrolithiasis are available to patients with the ultimate choice dependent on stone size, location, and patient factors. For over 30 years, the holmium: yttrium-aluminum-garnet (Ho:YAG) laser has been the gold standard for laser lithotripsy due to its efficiency in stone fragmentation irrespective of stone composition and its enviable safety profile. Different energies, pulse rates, pulse durations, and work settings are utilized based on stone density and surgeon intent for fragmentation versus dusting.

Basic physical principles underlie the effectiveness of the Ho:YAG laser, which made a revolution over two decades ago. Energy is transmitted through a flexible quartz fiber that varies in size from 150-1,000 micrometers making it amenable to flexible ureteroscopy. Its wavelength of 2,100 nm is effectively absorbed by water conferring a safety profile which is further bolstered by its 0.4mm depth of penetration. The photothermal mechanism by which it exerts force requires direct stone contact leading to stone vaporization. As a pulsed laser, holmium emits a cyclic burst of light wavelength with a corresponding omission. The average of the laser's pulses accounts for the power output. Contemporary advancements have led to utilization of higher power by taking advantage of the pulse technology. At present pulse duration can be lengthened from 350 microseconds to 1500 microseconds and utilized to reduce stone retropulsion. The latest evolution of the technology includes the aptly named "Moses Technology" (now in version 2.0) whereby a short vapor bubble precedes a longer duration, high energy pulse that can conserve energy by means of travel through the vapor bubble. This technology has been key in reducing stone retropulsion leading to improved ablation rates. Data has suggested that the Moses technology improves patient outcomes by reducing procedural duration and reducing fragmentation time.

A newer alternative to the Ho:YAG laser is the thulium fiber laser (TFL) lithotripter, introduced in 2018. It can provide greater power output from a smaller fiber core due to the diode construction with silica chemically doped with thulium ions. This is achieved by using a 50-150 micrometer optical laser fiber core rather than mirrors to focus light energy as in the Ho:YAG. Small form factor renders the fiber more adaptable in acute angle applications. The low power consumption of the TFL arises from fan cooling and plug efficiency permitting increased pulse repetition rates up to 2,000 - 2,200 Hz with pulse durations from 0.2 to 12 milliseconds. Due to these improvements, the TFL can both fragment and dust with moderated heat generation. Moreover, the TFL is compatible with variable operating room configurations based on its standard electrical wall socket (110V) making it more accessible. Similar to the Ho:YAG laser its wavelength varies between 1,908 and 1,940 nm bestowing a higher absorption coefficient in water which grants a similar safety profile owing to higher energy density focused at the tip of the laser fiber. In summation, the TFL has comparable results for stone ablation and low retropulsion with lower power consumption and less retropulsion leading to better dusting.

Recent studies have compared specific features of each laser to standardize best practices albeit with no clear winner. Pulse profiles differ with each laser. The Ho:YAG pulse has an acute spike in voltage with a dramatic drop within 150 microseconds whereas the TFL pulse profile has an acute upsurge that is sustained for the duration of the pulse. This inherent property within the TFL allows greater dialed in variability. With regard to energy absorption the TFL has been shown to be 4-5 times more effective thus correlating with lower pulsed energies for stone ablation in the in vitro setting. Lower pulsed energies in conjunction with increased pulse durations allow for less retropulsion with better dusting. The TFL has demonstrable improvements in stone free rates by more readily creating fine dust than can the Ho:YAG and the Ho:YAG-MOSES in in vivo settings. Not to be undone, the Ho:YAG laser has statistically higher ablation rates at slow speeds of 500 mm/min when using approximately identical energies and frequencies. Data suggests that higher ablation rates are more readily obtained at high-powered settings (24W) albeit with increased risk for thermal damage. Moreover, in vivo models suggest increased risk for urothelial tissue injury when using TFL in the absence or ureteral access sheaths owing to increased temperature within the collecting system. At best, current in vivo and in vitro studies lack certain corollary to clinical scenarios however they do suggest an equivalency for tissue temperature damage by either laser modality via high-power low-irrigation settings. When going head-to-head the Ho:YAG has shown superiority with denser calcium phosphate stones. TFL may confer greater stone clearance but has also been found to increase the rate of infectious complications. Other studies have concluded no significant clinical time advantage, stone free rate, complication, or patient related stone quality of life outcomes. Therefore as both lasers confer safety with effectiveness, surgeon preference and institutional preference may dictate technological approach.

Studies have begun to compare TFL to high power holmium with Moses technology for ureteroscopy and laser lithotripsy (URSLL), however, data is lacking as to the superior laser technology for medium or large stones approached antegrade in the mini percutaneous nephrolithotomy (PCNL) setting.

This is a single institution, single surgeon, randomized controlled trial that evaluates the holmium laser vs. the thulium laser for medium-to-large stones in the mini Percutaneous Nephrolithotomy setting. Patients will be screened and consented for participation in this study, and will be randomized to be treated using either the holmium or thulium laser for their procedure. This study aims to evaluate the efficiency of both FDA-approved lasers for this procedure to ascertain whether one of them has any advantage over the other. Procedural information will be evaluated as well as up to 90 day outcomes for the participants of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo mini PCNL for nephrolithiasis
* Stone burden (multiple stones acceptable) with largest stone 1cm - 3 cm in greatest dimension on bone window of noncontrast CT within a 6 month preoperative period.
* Able to give informed consent
* Age 21 or older

Exclusion Criteria:

* Patients scheduled to undergo concurrent non-PCNL procedure such as contralateral ureteroscopy
* Inability to give informed consent
* Age less than 21
* Body Mass Index (BMI) >45
* Pregnant or breastfeeding patients
* Stone burden outside of inclusion criteria range
* Untreated urinary tract infections
* Uncontrolled bleeding disorder and coagulopathy
* Abnormal upper tract anatomy such as presence of ureteral strictures or complete ureteropelvic junction (UPJ) obstruction
* Patients with urinary diversion such as ileal conduit or neobladder
* Any preexisting medical condition or situation that, in the investigator's opinion, could put the participant at significant risk, confound the study results, or interfere significantly with the participants' participation in the study
* Are currently prescribed buprenorphine or methadone, or carry active diagnosis of chronic opioid use disorder

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Laser Treatment Time | The duration of the procedure
  Measured in minutes and seconds. Total laser treatment time will be total cumulative lasing time.

SECONDARY OUTCOMES:
Retreatment rate | 90 days
  Participants undergoing ureteroscopy, shockwave lithotripsy or repeat percutaneous stone treatment for the same stone(s) within 90 days.
Total Operative Time | The duration of the operation
  The time the procedure takes, starting at time of instrument insertion after positioning and draping and end at instrument removal.
Stone-Free Rate | 8-12 weeks after surgery
  No fragments greater than 3 mm in greatest dimension measured on low-dose noncontrast CT imaging approximately 8-12 weeks after surgery.

OTHER OUTCOMES:
Length of stay | 0-72 hours following procedure
  Length of stay in hospital after procedure.
Safety Profile and Adverse Events | The duration of the operation and 90 days post procedure
  Loss of blood during the procedure, immediate and delayed complications, subsequent stone events, emergency department visits.
Subjective pain scores | Immediately postoperatively through stent removal (0-14 days)
  Mean and worst pain scores on the numerical rating scale (NRS) postoperatively and at time of discharge. Numerical rating scale is reported as integers 0-10, with 10 being the worst pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: David W Sobel, MD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sadiq AS, Atallah W, Khusid J, Gupta M. The Surgical Technique of Mini Percutaneous Nephrolithotomy. J Endourol. 2021 Sep;35(S2):S68-S74. doi: 10.1089/end.2020.1080. PMID 34499550
- [Background] Petzold R, Miernik A, Suarez-Ibarrola R. In Vitro Dusting Performance of a New Solid State Thulium Laser Compared to Holmium Laser Lithotripsy. J Endourol. 2021 Feb;35(2):221-225. doi: 10.1089/end.2020.0525. Epub 2020 Sep 9. PMID 32799650
- [Background] Jiang P, Okhunov Z, Afyouni AS, Ali S, Hosseini Sharifi SH, Bhatt R, Brevik A, Ayad M, Larson K, Osann K, Patel RM, Landman J, Clayman RV. Comparison of Superpulse Thulium Fiber Laser vs Holmium Laser for Ablation of Renal Calculi in an In Vivo Porcine Model. J Endourol. 2023 Mar;37(3):335-340. doi: 10.1089/end.2022.0445. PMID 36401505
- [Background] Martov AG, Ergakov DV, Guseynov M, Andronov AS, Plekhanova OA. Clinical Comparison of Super Pulse Thulium Fiber Laser and High-Power Holmium Laser for Ureteral Stone Management. J Endourol. 2021 Jun;35(6):795-800. doi: 10.1089/end.2020.0581. Epub 2021 Jan 13. PMID 33238763
- [Background] Soto-Palou F, Chen J, Medairos R, Zhong P, Antonelli J, Preminger GM, Lipkin ME. In Pursuit of the Optimal Dusting Settings with the Thulium Fiber Laser: An In Vitro Assessment. J Endourol. 2023 Aug;37(8):914-920. doi: 10.1089/end.2023.0168. Epub 2023 Jun 26. PMID 37300481
- [Background] Matlaga BR, Chew B, Eisner B, Humphreys M, Knudsen B, Krambeck A, Lange D, Lipkin M, Miller NL, Monga M, Pais V, Sur RL, Shah O. Ureteroscopic Laser Lithotripsy: A Review of Dusting vs Fragmentation with Extraction. J Endourol. 2018 Jan;32(1):1-6. doi: 10.1089/end.2017.0641. Epub 2017 Nov 27. PMID 29061070
- [Background] Kronenberg P, Traxer O. The laser of the future: reality and expectations about the new thulium fiber laser-a systematic review. Transl Androl Urol. 2019 Sep;8(Suppl 4):S398-S417. doi: 10.21037/tau.2019.08.01. PMID 31656746
- [Background] Darr C, Krafft U, Panic A, Tschirdewahn S, Hadaschik BA, Rehme C. Renal duplication with ureter duplex not following Meyer-Weigert-Rule with development of a megaureter of the lower ureteral segment due to distal stenosis - A case report. Urol Case Rep. 2019 Nov 14;28:101038. doi: 10.1016/j.eucr.2019.101038. eCollection 2020 Jan. PMID 31763165
- [Background] Nikoufar P, Hodhod A, Fathy M, Zakaria AS, Shabana W, Abdul Hadi R, Abdelkawi IF, Alaradi H, Abbas L, Alaref A, Shahrour W, Elmansy H. Thulium Fiber Laser vs Pulse-Modulated Holmium MOSES Laser in Flexible Ureteroscopy for the Management of Kidney Stones: A Single-Center Retrospective Analysis. J Endourol. 2023 Oct;37(10):1081-1087. doi: 10.1089/end.2023.0284. Epub 2023 Sep 20. PMID 37597211
- [Background] Ibrahim A, Elhilali MM, Fahmy N, Carrier S, Andonian S. Double-Blinded Prospective Randomized Clinical Trial Comparing Regular and Moses Modes of Holmium Laser Lithotripsy. J Endourol. 2020 May;34(5):624-628. doi: 10.1089/end.2019.0695. Epub 2020 Apr 3. PMID 32143552
- [Background] Okhunov Z, Jiang P, Afyouni AS, Ayad M, Arada R, Brevik A, Akopian G, Patel RM, Landman J, Clayman RV. Caveat Emptor: The Heat Is "ON"-An In Vivo Evaluation of the Thulium Fiber Laser and Temperature Changes in the Porcine Kidney During Dusting and Fragmentation Modes. J Endourol. 2021 Nov;35(11):1716-1722. doi: 10.1089/end.2021.0206. Epub 2021 Oct 18. PMID 33906433
- [Background] Jiang P, Peta A, Brevik A, Arada RB, Ayad M, Afyouni AS, Limfueco L, Nguyen N, Palma A, Patel RM, Landman J, Clayman RV. Ex Vivo Renal Stone Dusting: Impact of Laser Modality, Ureteral Access Sheath, and Suction on Total Stone Clearance. J Endourol. 2022 Apr;36(4):499-507. doi: 10.1089/end.2021.0544. PMID 34693735
- [Background] Sierra A, Corrales M, Kolvatzis M, Panthier F, Pinero A, Traxer O. Thermal Injury and Laser Efficiency with Holmium YAG and Thulium Fiber Laser-An In Vitro Study. J Endourol. 2022 Dec;36(12):1599-1606. doi: 10.1089/end.2022.0216. PMID 35793107
- [Background] Petzold R, Suarez-Ibarrola R, Miernik A. Temperature Assessment of a Novel Pulsed Thulium Solid-State Laser Compared with a Holmium:Yttrium-Aluminum-Garnet Laser. J Endourol. 2021 Jun;35(6):853-859. doi: 10.1089/end.2020.0803. Epub 2020 Dec 3. PMID 33191783
- [Background] Castellani D, Fong KY, Lim EJ, Chew BH, Tailly T, Emiliani E, Teoh JY, Chai CA, Heng CT, Ong Lay Keat W, Tanidir Y, Ragoori D, Galosi AB, Singh A, Bin Hamri S, Traxer O, Somani BK, Gauhar V. Comparison Between Holmium:YAG Laser with MOSES Technology vs Thulium Fiber Laser Lithotripsy in Retrograde Intrarenal Surgery for Kidney Stones in Adults: A Propensity Score-matched Analysis From the FLEXible Ureteroscopy Outcomes Registry. J Urol. 2023 Aug;210(2):323-330. doi: 10.1097/JU.0000000000003504. Epub 2023 May 1. PMID 37126223
- [Background] Haas CR, Knoedler MA, Li S, Gralnek DR, Best SL, Penniston KL, Nakada SY. Pulse-modulated Holmium:YAG Laser vs the Thulium Fiber Laser for Renal and Ureteral Stones: A Single-center Prospective Randomized Clinical Trial. J Urol. 2023 Feb;209(2):374-383. doi: 10.1097/JU.0000000000003050. Epub 2023 Jan 9. PMID 36621994
- [Background] Mahajan AD, Mahajan SA. Thulium fiber laser versus holmium:yttrium aluminum garnet laser for stone lithotripsy during mini-percutaneous nephrolithotomy: A prospective randomized trial. Indian J Urol. 2022 Jan-Mar;38(1):42-47. doi: 10.4103/iju.iju_331_21. Epub 2022 Jan 1. PMID 35136294
- [Background] Patil A, Reddy N, Shah D, Singh A, Ganpule A, Sabnis R, Desai M. High-Power Holmium with MOSES Technology or Thulium Fiber Laser in MiniPerc with Suction: A New Curiosity. J Endourol. 2022 Oct;36(10):1348-1354. doi: 10.1089/end.2021.0915. Epub 2022 Aug 17. PMID 35331003
- [Background] Cella D, Choi SW, Condon DM, Schalet B, Hays RD, Rothrock NE, Yount S, Cook KF, Gershon RC, Amtmann D, DeWalt DA, Pilkonis PA, Stone AA, Weinfurt K, Reeve BB. PROMIS(R) Adult Health Profiles: Efficient Short-Form Measures of Seven Health Domains. Value Health. 2019 May;22(5):537-544. doi: 10.1016/j.jval.2019.02.004. PMID 31104731
- [Background] Higgins AM, Ganesan V, Ghani KR, Agarwal DK, Borofsky MS, Dauw CA. The 2023 Stone-Free CT Mandate: Addressing the Two Sides of the Debate. J Endourol. 2022 Dec;36(12):1522-1525. doi: 10.1089/end.2022.0610. Epub 2022 Nov 7. PMID 36150029
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- See also: Holmium Laser — https://www.bostonscientific.com/en-US/medical-specialties/urology/products/moses-technology.html
- See also: Thulium Laser — https://medical.olympusamerica.com/products/soltive%E2%84%A2-superpulsed-laser-system

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT06266793/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT06266793/ICF_001.pdf